CLINICAL TRIAL: NCT05873023
Title: Effect of Chewing Gum on Cognitive Function
Brief Title: Chewing Gum and Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Collaborators: Bobath Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202105034
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group chew one unscented gum provided by the study for 12 weeks. The participants are instructed to masticate a gum for 20 minutes every day, alternately for 10 minutes on the right side and 10 minutes on the left side.
  After chewing gum, they perform masticatory muscle stretching and tongue exercises. After they finish chewing the gum, he or she reports completion by posting a proof photo in the KakaoTalk chat room.
  Interventions: Other: Chewing gum
- Control (No Intervention): The control group does not participate in chewing gum.

INTERVENTIONS:
Other: Chewing gum — chewing gum everyday for 12 weeks. Alternate chewing for 10 minutes on the right and 10 minutes on the left.
  Arms: Intervention

SUMMARY:
This study is to investigate whether the improvement or maintenance of cognitive function is superior to the control group when gum chewing is performed in elderly people with subjective cognitive decline or mild cognitive impairment.

DETAILED DESCRIPTION:
The intervention group chew one unscented gum provided by the study for 12 weeks. Using KakaoTalk, the coordinator sends a chewing gum alarm.

The participants are instructed to masticate a gum for 20 minutes every day, alternately for 10 minutes on the right side and 10 minutes on the left side.

After chewing gum, they perform masticatory muscle stretching and tongue exercises. After they finish chewing the gum, he or she reports completion by posting an authentication photo in the KakaoTalk chat room.

The research coordinator checks the certification on a weekly basis and sends a separate phone call to encourage participants who do not chew gum more than twice a week.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 79 years of age
* All posterior teeth are evenly occluded on both sides, and those who have lost 4 or less teeth in the posterior teeth
* Those who scored 50 points or less on the periodontal disease self-checklist
* Meet the diagnostic criteria for subjective cognitive decline or mild cognitive impairment
* Provide written informed consent

Exclusion Criteria:

* Those who have difficulty in chewing due to toothache, periodontal disease, temporomandibular joint disease, severe malocclusion, shaking teeth, etc.
* Those who wear dentures on the upper or lower teeth
* Dementia
* Major psychiatric illness such as major depressive disorders
* Other neurodegenerative disease (e.g., Parkinson's disease)
* Other serious or unstable medical disease such as acute or severe asthma, active gastric ulcer, severe liver disease, or severe renal disease, or any medical conditions preventing to complete the study as judged by the study physician
* Severe loss of vision, hearing, or communicative disability
* Significant laboratory abnormality that may result in cognitive impairment
* Any conditions preventing cooperation as judged by the study physician
* Coincident participation in any other intervention trial
* Those who are planning dental treatment such as preservation, prosthetics, and implants during the research period

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Change of cognition | Change from Baseline at 12 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status (range 40-160). Higher scores indicate better performance.

SECONDARY OUTCOMES:
Change of global cognition | Change from Baseline at 12 weeks
  Korean Mini-Mental State Examination-2 (range, 0-30). Higher scores indicate better performance.
Change of function | Change from Baseline at 12 weeks
  Clinical Dementia Rating scale-Sum of Boxes (range 0-18). Higher scores indicate worse performance.
Change of depression | Change from Baseline at 12 weeks
  Geriatric Depression Scale-15 items (range 0-15). Higher scores indicate worse mood.
Change of activities of daily living | Change from Baseline at 12 weeks
  Bayer Activities of Daily Living (range 1-10). Higher scores indicate worse performance.
Change of quality of life | Change from Baseline at 12 weeks
  Quality of life-Alzheimer's disease (range 0-52). Higher scores indicate better performance.

OTHER OUTCOMES:
Change of cortical thickness and brain network function | Change from Baseline at 12 weeks
  brain MRI (3D-T1 weighted images and resting state functional MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Hae Ri Na, MD, PhD, Principal Investigator — Bobath Memorial Hospital
Locations (4):
- South Korea (4):
  - Bobath Memorial Hospital, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Ewha Womans Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available for 2 years since March 2025.
Access Criteria: Reasonable request